CLINICAL TRIAL: NCT06066853
Title: Hyperscan Neuroimaging to Reveal the Brain Mechanisms Supporting Analgesia Following MDMA-assisted Therapy for Fibromyalgia
Brief Title: MDMA-assisted Therapy for Fibromyalgia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Multidisciplinary Association for Psychedelic Studies (Other)
Responsible Party: Principal Investigator, Vitaly Napadow, LICAC, PhD, Professor, Harvard Medical School, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P002488
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Fibromyalgia
Keywords: N-Methyl-3,4-methylenedioxyamphetamine; Fibromyalgia; MDMA; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Single arm open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: MDMA — MDMA-assisted psychotherapy

SUMMARY:
Fibromyalgia is a debilitating chronic pain disorder. Based on prior research with MDMA, it can be hypothesized MDMA-assisted therapy in fibromyalgia patients may increase the range of positive emotions, interpersonal trust, and heighten the state of empathic rapport that can lead to an enhanced patient-clinician interaction and to initiate reattribution processes targeting dysfunctional thoughts towards pain. Therapeutic alliance, i.e. a positive patient-clinician relationship, is already acknowledged as an essential component for MDMA-assisted therapy. Despite its importance, the patient-clinician interaction and the neuroscience supporting patient/clinician therapeutic alliance has received almost no attention in MDMA research. The investigators will examine the potential therapeutic benefit of MDMA-assisted therapy for fibromyalgia. Additionally, this study will also target secondary objectives including the investigation of the clinical and physiological response (i.e. brain-to-brain concordance) supporting enhanced patient-clinician therapeutic alliance in fibromyalgia patients. The study includes two Experimental Sessions of therapy with MDMA combined with neuroimaging, along integrative therapy, baseline neuroimaging, and a 3 month follow up.

DETAILED DESCRIPTION:
If the participant agrees to engage in this research study, they will be asked to complete the following study visits:

Screening (Visit 1):

At this visit the participant will review and sign the consent form. If informed consent is given, the investigators will proceed to screening. During screening, the study personnel will decide if eligibility criteria are met. The study staff will ask about medical and psychiatric history, medications, and any other conditions. They will then further assess eligibility through clinical lab tests, a drug screen, and pregnancy test for those able to become pregnant. The drug screen will include at minimum: amphetamines, barbiturates, cocaine, opioids, cannabinoids, and benzodiazepines. Participants will also complete a symptom-directed physical exam and vitals (blood pressure, temperature, and respiratory and heart rate) will be assessed. An electrocardiogram (ECG), a test that measures the rhythm and rate of the heart, will be performed. Additional cardiovascular evaluation and risk mitigation will be completed to determine eligibility if the participant has cardiac risk factors, but no other evidence of significant cardiovascular or cerebrovascular disease.

At the screening visit study staff will measure the participant's responses to pressure pain, using an inflatable cuff that is placed on the lower leg. Different pressure intensities to inflate the cuff will be used. The participant will be asked to complete several questionnaires that will assess personality and other traits along with questionnaires to assess pain. Participants found eligible after the screening visit will be enrolled in the study.

All participants are required to identify a support person. This person will be responsible for staying with the participant on the evenings of the experimental sessions and will meet with the therapy team to receive training regarding their role. All participants will also be required to identify an escort, who will accompany the participant to and from the study site for each experimental session. This may be the same person as the support person, or it may be someone else.

Baseline EEG and MRI (Visits 2 and 3):

Following enrollment, participants will complete a baseline electroencephalography (EEG) scan followed by a functional magnetic resonance imaging (fMRI) scan. At the EEG scan participants will be asked to view and reflect on various statements and to complete a cuff pressure task, in which they will receive various cuff pressures to their left leg. While participants are doing these tasks, the activity of the brain will be monitored using EEG and vitals will be measured.

At the fMRI scan participants will be asked to change out of their clothes and into an MRI-compatible hospital gown and pants to ensure safety. They will be asked to remove any metal objects including jewelry, any piercings, and hair pins. Participants will be given earplugs to reduce the loud noises of the MRI machine. Participants will be able to communicate with the study doctors and MRI staff during the procedures. While in the scanner, participants will complete the same tasks as described in the EEG session. The clinician will be positioned in a different scanner, and video transfer between the two scanners will enable the patient and clinician to view one another's face on a screen for some of the tasks.

In order to quality check the interaction between the patient and the clinician, parts of these scans will be recorded on a videotape.

Preparatory Period (Visits 4-6):

Following baseline scans, participants will undergo three weekly preparatory sessions, with each session lasting about 90 minutes. During these visits participants will meet with their therapy team to learn more about fibromyalgia and develop rapport with their clinicians. The therapy team will help prepare participants for the experimental visits. During this period, participants will undergo medication tapering if necessary. Prior to the final preparatory session, the investigators will do a final assessment of eligibility and confirm that all medication tapering is complete.

Experimental Period (Visits 7-12):

The experimental period will consist of two MDMA-assisted therapy sessions and four integrative sessions. Each of the experimental sessions will last for about 8 hours. At the beginning of the experimental sessions, participants will complete a symptom-directed physical exam, a urine drug screen, and a pregnancy test if applicable. These tests must be negative for the visit to proceed. Participants will be asked to confirm they have not consumed nicotine or caffeine for the past 2 hours and have not consumed food for the past 10 hours. They will complete several questionnaires and will have a quick interview with the therapy team to discuss goals, intentions, and concerns related to the MDMA-assisted therapy session. Vitals will be recorded just before drug administration.

Participants will receive an initial dose of 100 mg of MDMA. They will swallow capsules of study drug with water under the supervision of study staff. The participant will sit or recline on comfortable furnishings and complete MDMA-assisted therapy with their clinicians. A supplemental dose of 50 mg of study drug will be administered 1.5 to 2 hours after the initial dose as seen fit by the therapy team.

About three hours post initial drug administration participants will have an EEG (Visit 7) or fMRI (Visit 10) scan. Throughout these scans participants will remain in contact with their therapy team. These scans will be include the same tasks and procedures as the baseline scans. Following the EEG or fMRI scan, participants will remain with the therapy team until the study drug effects have subsided, their vitals are stable, and their support person or escort has arrived.

Following each experimental visit there will be two integrative sessions, which will consist of 90 minutes of therapy. At these visits participants will discuss and review events from the experimental session. One of the integrative visits (Visit 11) will include an EEG scan during the therapy session.

Follow-up (Visit 13):

About four weeks after the final integration session, participants will be asked to complete a virtual follow-up visit to complete a short interview and answer some final questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 21 years to 65 years of age inclusive, at the time of signing the informed consent.
* Have a clinical diagnosis of fibromyalgia and meet the Wolfe et al 2011 research criteria for fibromyalgia for at least one year.
* Typical fibromyalgia pain intensity of 4/10 or greater.
* Fluent in speaking and reading English.
* Able to swallow pills.
* Agree to have some study visits audiovisually recorded, including Experimental Sessions/ neuroimaging sessions.
* Able to provide a contact (relative, spouse, close friend, or other support person) who is willing and able to be reached by the investigators in the event of the participant becoming unwell or unreachable.
* Able to identify appropriate support person(s) to stay with the participant on the evenings of the Experimental Sessions
* Have a body weight of at least 45 kilograms (kg). Participants with a body weight of 45 to 48 kg must also have a body mass index (BMI) within the range of 18 to 30 kg/m2
* Participants assigned female sex at birth must not be pregnant or become pregnant throughout participation in the study
* Capable of giving signed informed consent
* Are on stable doses of allowable medication for 30 days prior to entering the study and agree not to change medications or dosages during the trial, except for medications falling under the tapering scheduling

Exclusion Criteria:

* Presence of any medical or psychiatric illness that is judged to interfere with the study (ex. Fibromyalgia, PTSD, bipolar, schizophrenia) determined by a self-report measure.
* Presence of any contraindications to fMRI scanning or EEG scanning. (ex. Cardiac pacemaker, metal implants, fear of enclosed spaces, pregnancy).
* Unwillingness to receive brief experimental pain
* Lower extremity pain or vascular issues that may interfere with the study procedures
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Have a history of any medical condition that could make receiving a sympathomimetic drug harmful because of increases in blood pressure and heart rate. This includes, but is not limited to, a history of myocardial infarction, cerebrovascular accident, heart failure, severe coronary artery disease, or aneurysm.
* Have a diagnosis of uncontrolled hypertension, defined as repeated blood pressure readings of ≥140 mmHg systolic or ≥90 mmHg diastolic.
* Have a history of ventricular arrhythmia at any time, other than occasional premature ventricular contractions (PVCs) in the absence of ischemic heart disease.
* Have Wolff-Parkinson-White syndrome or any other accessory pathway that has not been successfully eliminated by ablation.
* Have a history of arrhythmia, other than premature atrial contractions (PACs) or occasional PVCs in the absence of ischemic heart disease, within 12 months of screening.
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
* Have engaged in a new form of psychiatric or mental health care within 12 weeks of enrollment, including Electroconvulsive Therapy (ECT), and ketamine-assisted therapy.
* Have a current moderate or severe alcohol or cannabis use disorder within the 12 months prior to enrollment.
* Have an active illicit drug (other than cannabis) or prescription drug substance use disorder at any severity within 12 months prior to enrollment.
* Any participant presenting current serious suicide risk, as determined through psychiatric interview, responses to C-SSRS, and clinical judgment of the investigator will be excluded; however, history of suicide attempts is not an exclusion.
* Unable or unwilling to safely taper-off prohibited psychiatric and non-psychiatric medication with exceptions determined by study staff or require use of prohibited medications during experimental sessions.
* Require use of concomitant medications that could prolong the QT interval during Experimental Sessions.
* Have used Ecstasy (unregulated material represented as containing MDMA) more than 10 times within the last 10 years, or at least once within 6 months of the first Experimental Session.
* Current enrollment in any other clinical study involving an investigational study treatment or any other type of medical research, unless approved by the study clinician.
* Have current Personality and/or Psychotic Disorders.
* Have a current eating disorder with compensatory behaviors.
* Have current major depressive disorder with psychotic features.
* Have a history of, or a current primary psychotic disorder, bipolar affective disorder type 1.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the sponsor-investigator or study clinician, contraindicates participation in the study.
* Are currently engaged in compensation litigation whereby financial gain would be achieved from prolonged symptoms of fibromyalgia or any psychiatric disorders.
* Lack social support or lack a stable living situation.
* Previous participation in a MAPS-sponsored MDMA clinical trial.
* Employees (and their immediate family members) of MAPS, MAPS Public Benefit Corporation, or MAPS Europe B.V; or individuals in a personal relationship with the site investigator.
* Presence of any medical or psychiatric illness that is judged to interfere with trial
* Presence of any contraindications to fMRI scanning or EEG scanning (ex. Cardiac pacemaker, metal implants, fear of closed spaces)
* Lower extremity pain or vascular issues that may interfere with study procedures
* Comorbid chronic pain condition that is rated by the subject as more painful than fibromyalgia
* Have any severe anxiety disorders or significant anxiety symptoms interfering with fMRI scanning (e.g. panic)
* Is a current patient of the matched dyad clinician enrolled in the study
* Would present a serious risk to others as established through clinical interview and contact with treating psychiatrist.
* Have any current problem which, in the opinion of the sponsor-investigator or study clinician, might interfere with study participation or prevent satisfactory completion of study protocol.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported pain severity and pain interference (Brief Pain Inventory) | BPI will be assessed at five timepoints (Visits 1, 7, 10, 12, and 13) throughout the study, spanning approximately 3 months.
  Brief Pain Inventory (BPI) is a validated 16 item questionnaire designed to assess the severity and interference of pain experienced. Pain severity is assessed on a scale from 0 (no pain) to 10 (severe pain). Pain interference is assessed on a scale from 0 (no interference) to 10 (severe interference).

CONTACTS AND LOCATIONS:
Overall Officials: Vitaly Napadow, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No